CLINICAL TRIAL: NCT03219827
Title: Pilot Study: Characterization of the Immune Phenotype of Patients Allergic to Wasp Venom or Penicillin
Acronym: WasPenIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-036
Record Dates: First submitted 2017-06-16; First posted 2017-07-18 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients allergic to wasp venom (Experimental): Patient with major allergic reaction to wasp venom.
  * Blood samples collection at visit 1, at visit 2 (4 weeks after visit 1), at visit 3 (one year after treatment onset)
  * After visit 1, an allergen-specific immunotherapy will be conducted as part of the classical patient care program.
  Interventions: Other: Human biological samples
- Patients allergic to penicillin (Experimental): Patient with major allergic reaction to penicillin.
  - Blood samples collection at visit 1 and at visit 2 (4 weeks after visit 1= end of study, none treatment will be evaluated in this arm)
  Interventions: Other: Human biological samples

INTERVENTIONS:
Other: Human biological samples — Blood samples collection

SUMMARY:
Severity of allergic reactions are highly variable from one individual to another, they can range from absent to life threatening. Allergic manifestations and specifically those of anaphylactic reactions are generally attributed to an IgE-dependent activation of mast cells and/or basophils followed by the release of histamine. Recently however evidence accumulated that other pathways might similarly contribute or even trigger anaphylaxis. Moreover, while the variance in human populations is an important subject to scientific research, medical practices and public health policies typically take a 'one for all' approach to disease management and drug development. Indeed, individual heterogeneity in the immune response can have a big impact on the likelihood to respond to therapy. Because of the complexity of immune responses in the individual and within the population, it has not been possible thus far to define the parameters (genetic or environmental) that define the immune system of allergic patients and its natural occurring variability. Thanks to the efforts that have been made in the framework of the Labex "Milieu Intérieur" study genetic, immunological and environmental factors have been identified that can be linked to the heterogeneity of immune responses in healthy individuals. By comparing these already available data from healthy individuals to a novel cohort of patients with defined severe allergic manifestations, we will be able to identify for the first time immunological and environmental parameters that are common to patients with severe allergies and identify those parameters that distinguish allergic patients from the healthy donor cohort. This analysis will thus open new perspectives on deregulated immune pathways in allergic patients allowing to orient future treatment approaches. Furthermore, comparing immune responses before and after allergen-specific immunotherapy will help understanding, which changes in immune responses are causal to a successful treatment. Importantly, this analysis will shed light on the individual differences that may predict the outcome of treatment approaches and propose novel markers of its success.

DETAILED DESCRIPTION:
Severity of allergic reactions are highly variable from one individual to another, they can range from absent to life threatening. Allergic manifestations and specifically those of anaphylactic reactions are generally attributed to an IgE-dependent activation of mast cells and/or basophils followed by the release of histamine. Recently however evidence accumulated that other pathways might similarly contribute or even trigger anaphylaxis. Moreover, while the variance in human populations is an important subject to scientific research, medical practices and public health policies typically take a 'one for all' approach to disease management and drug development. Indeed, individual heterogeneity in the immune response can have a big impact on the likelihood to respond to therapy. Because of the complexity of immune responses in the individual and within the population, it has not been possible thus far to define the parameters (genetic or environmental) that define the immune system of allergic patients and its natural occurring variability. Thanks to the efforts that have been made in the framework of the Labex "Milieu Intérieur" study genetic, immunological and environmental factors have been identified that can be linked to the heterogeneity of immune responses in healthy individuals. By comparing these already available data to a novel cohort of patients with defined severe allergic manifestations, we will be able to identify for the first time immunological and environmental parameters that are common to patients with severe allergies and identify those parameters that distinguish allergic patients from the healthy donor cohort. This analysis will thus open new perspectives on deregulated immune pathways in allergic patients allowing to orient future treatment approaches. Furthermore, comparing immune responses before and after allergen-specific immunotherapy will help understanding, which changes in immune responses are causal to a successful treatment. Importantly, this analysis will shed light on the individual differences that may predict the outcome of treatment approaches and propose novel markers of its success. Hence, it will give important insights for the individually adapted treatment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Allergic subjects having done either an allergic reaction at least of grade 3 according to Müller1 or a quincke edema in response to a wasp sting or penicillin intake, otherwise considered as healthy by the investigator based on medical history, clinical examination and laboratory results (blood sampling for laboratory assessments should be done at V0 and only after signed informed consent).
* Subjects who, according to the investigator, can and will comply with the requirements of the protocol and are available for all scheduled visits at the investigational site.
* Wasp or penicillin allergic but otherwise healthy male and female aged between 20 and 69 years.
* 18.5 <= BMI >= 32 kg/m2
* Ability to give their consent in writing
* Must understand spoken and written French
* Affiliated to the French social security or assimilated regimes

Exclusion Criteria:

* Subjects who cannot participate according to their status on the registry mentioned at Art L.1121-16 of the French Public Health Code
* Participation in another Clinical study in the last 3 months in which the subject has been exposed to an investigational product (pharmaceutical product or placebo or medical device) or concurrent participation in another clinical study during the study period
* Travel in (sub-)tropical countries within the last 3 months
* For women: pregnant or breastfeeding or intending to become pregnant or peri-menopausal
* Any physical exercise within the last 8 hours before inclusion (V1) and before (V2)
* Presence of evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential patient unable/unlikely to participate in the study satisfactorily.
* Severe/chronic/recurrent pathological conditions,
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the V0, V1 or V2. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
* Chronic administration of NSAIDs, including aspirin: prolonged intake (> 2 weeks) within 6 months before [exception for low dose aspirin: maximum 250mg/daily, see 5.1]
* Receipt of any vaccination 3 months before the inclusion or planning to receive any vaccination during the study
* Receipt of blood products or immunoglobulins within 3 months prior the inclusion or planning to receive blood products or immunoglobulins during the study
* Hemoglobin measurement less than 10.0 g/dL for women and less than 11.5 g/dL for men
* Platelet count less than 120.000/mm3
* ALAT and/or ASAT > 3 times the upper limit of the norm (ULN)

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Immune phenotype of allergic patients | 3 years
  Determination of the immune phenotype of allergic patients through flow cytometric analysis of major blood cell populations
Immune phenotype of allergic patients by determination of cytokine/chemokine levels | 3 years
  Measurement of cytokine/chemokine levels in whole bood following stimulation with 6 immune stimulators.

SECONDARY OUTCOMES:
Differences in immune responses before and after immunotherapy measured by flow cytometric analysis. | 3 years
  Differences between immune responses between patients before and after allergic -specific immunotherapy and between cured and non-cured patients measured by flow cytometric analysis
Differences in immune responses before and after immunotherapy | 3 years
  Differences between immune responses between patients before and after allergic -specific immunotherapy and between cured and non-cured patients measured by cytokine/chemokine levels in whole bood following stimulation with 6 immune stimulators.
Antibody repertoire determination measured by antigen specific ELISA. | 3 years
  Antibody repertoire in wasp venom allergic patients before and after allergen-specific immunotherapy. To determine changes in antigen recognition and subclass composition we will perform antigen specific ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Seringulian, Principal Investigator — Hôpital Saint Joseph
Locations (2):
- France (2):
  - Hôpital Saint Joseph, Paris
  - Service de Pneumologie Hôpital Bichat, Paris

IPD SHARING:
Plan to Share IPD: No